CLINICAL TRIAL: NCT02726321
Title: Early Detection of Subclinical Carotid Atherosclerosis Through Autonomic Testing
Brief Title: Autonomic Testing in Subclinical Carotid Atherosclerosis
Acronym: AtheroDetect
Status: Completed | Type: Observational
Sponsor: Universidade Camilo Castelo Branco (Other)
Responsible Party: Principal Investigator, Ovidiu Constantin Baltatu, Professor, Universidade Camilo Castelo Branco
Other Study IDs: BR-003-SJC
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2016-03

CONDITIONS: Subclinical Carotid Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Atherosclerotic carotid intima-media thickness (IMT) may be associated with alterations in the sensitivity of carotid and subclavian baroreceptors.

Aim: The aim of this study is to investigate if carotid IMT is associated with changes in the autonomic modulation of the heart rate variability (HRV).

Methods: This is a prospective cross-sectional study. The carotid IMT is determined by B-mode and duplex ultrasonography. The cardiovagal function was determined through linear and nonlinear measures of HRV. Linear regression models, adjusted for demographics, comorbidities, body mass index, waist-hip-ratio, and left ventricular ejection fraction will be used to evaluate the association between HRV parameters and carotid IMT.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic patients aged 18 years and older without a history of transient ischemic attack, stroke, or other neurologic signs or symptoms are selected to participate in the study.

Exclusion Criteria:

* Patients with symptomatic carotid artery stenosis were excluded if the patient had transient or permanent focal neurologic symptoms related to the ipsilateral retina or the cerebral hemisphere.
* Patients with heart rhythm disorders, pacemaker, heart failure, ejection fraction less than 0.45, chronic renal failure on hemodialysis, severe liver failure, myocardial infarction, endarterectomy, carotid angioplasty, carotid dissection and carotid occlusion were excluded.
* Patients receiving drugs known to interfere with autonomic function, such as beta-blockers, calcium channel blockers, angiotensin-converting enzyme inhibitors, vasodilators, statins, neuroleptics and nasal vasoconstrictors, were discontinued for 24 hours before the tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred to the Heart Institute of Santa Casa Charity (IACOR), Fernandopolis, Brazil for noninvasive carotid artery duplex ultrasonography. Carotid arteriosclerotic disease is evaluated through measuring the IMT and calculating the plaque score.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
carotid intima-media thickness (IMT) | 1 day
  carotid IMT is determined by B-mode and duplex ultrasonography
cardiovagal function | 1 day
  the cardiovagal function is determined through linear and nonlinear measures of HRV

CONTACTS AND LOCATIONS:
Overall Officials: Ovidiu C Baltatu, MD PhD, Study Chair — Universidade Camilo Castelo Branco; Valter L Pereira Jr., MD, Study Director — Heart Institute of Santa Casa Charity (IACOR) Fernandopolis

IPD SHARING:
Plan to Share IPD: No